CLINICAL TRIAL: NCT03291145
Title: Exploring Mechanisms and Morphology of QT Interval Prolongation - An Inheritable as Well as an Inducible Phenomenon
Brief Title: Exploring Mechanisms and Morphology of QT Interval Prolongation
Acronym: TriQarr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Peter Marstrand, Medical Doctor, Research Fellow, Herlev and Gentofte Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 260910000001
Record Dates: First submitted 2017-08-14; First posted 2017-09-25 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Long Qt Syndrome 1-2; Sudden Cardiac Death
Keywords: Long QT Syndrome
MeSH Terms: conditions — Long Qt Syndrome 1-2; Death, Sudden, Cardiac; Long QT Syndrome | interventions — Adrenergic beta-Antagonists; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta Blockers (Experimental): With and without Beta Blockers
  Interventions: Drug: Beta Blockers
- Spironolactone (Experimental): With and without Spironolactone
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Beta Blockers — With and without Beta Blockers
  Arms: Beta Blockers
Drug: Spironolactone — Brisk Standing before and after seven days treatment with Spironolactone
  Arms: Spironolactone

SUMMARY:
The projects will try and optimise the risk stratification for patients with Long QT syndrome by investigating how the exposure of physical and acoustic stress will affect the QT-dynamics and if beta blockers protect against arrhythmias by suppressing this dynamic QT-prolongation. Furthermore, the project will investigate the effects of Spironolactone on the QT-dynamics tested by "Brisk Standing".

First, patients are tested with known arrhythmic triggers and they are then administered thier normal dose of beta blockers. Hereafter, "Brisk Standing" test is performed and the patients are on Spironolactone for seven days. After seven days treatment the "Brisk Standing" is repeated.

DETAILED DESCRIPTION:
The aim of the projects is to try and optimise the risk stratification for patients with Long QT syndrome by investigating how the exposure of physical and acoustic stress will affect the QT-dynamics and if beta blockers protect against arrhythmias by suppressing this dynamic QT-prolongation. Furthermore, the project will investigate the effects of Spironolactone on the QT-dynamics tested by "Brisk Standing".

First, patients are tested with known arrhythmic triggers and they are then administered thier normal dose of beta blockers. Hereafter, "Brisk Standing" test is performed and the patients are on Spironolactone for seven days. After seven days treatment the "Brisk Standing" is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Verified Long QT syndrome mutation, subtype 1 or 2.
* over 18 years of age

Exclusion Criteria:

* Atrioventricular block,
* Left bundle branch block,
* Left ventricular hypertrophy,
* Pace rhythm,
* ST-deviations >1 mm),
* Left ventricular ejection fraction <50 % and significant valvulopathy,
* Unstable psychiatric disease
* Unstable cardiovascular disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
QTc | 7 days
  Corrected QT

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Herlev, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marstrand P, Almatlouh K, Kanters JK, Graff C, Christensen AH, Bundgaard H, Theilade J. Effect of moderate potassium-elevating treatment in long QT syndrome: the TriQarr Potassium Study. Open Heart. 2021 Sep;8(2):e001670. doi: 10.1136/openhrt-2021-001670. PMID 34531279
- [Derived] Marstrand P, Almatlouh K, Kanters JK, Graff C, Christensen AH, Bundgaard H, Theilade J. Long QT syndrome type 1 and 2 patients respond differently to arrhythmic triggers: The TriQarr in vivo study. Heart Rhythm. 2021 Feb;18(2):241-249. doi: 10.1016/j.hrthm.2020.08.017. Epub 2020 Aug 31. PMID 32882399